CLINICAL TRIAL: NCT02595567
Title: Indwelling Tunneled Catheter Placement for Treatment of Hepatic Hydrothorax
Brief Title: Catheter Placement for Hepatic Hydrothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Alexander Chen, Director Interventional Pulmonolgy, Assistant Professor of Medicine, Division of Pulmonary & Critical Care, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108320
Record Dates: First submitted 2015-09-01; First posted 2015-11-03 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Pleural Effusion
Keywords: Liver disease; Pleural effusion
MeSH Terms: conditions — Pleural Effusion; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITPC (Other)
  Interventions: Device: Indwelling tunneled pleural catheter (ITPC)

INTERVENTIONS:
Device: Indwelling tunneled pleural catheter (ITPC) — ITPCs have been shown to successfully and safely control dyspnea in patients with malignant pleural effusions. Compared to the large amount of published data regarding the use of indwelling tunneled pleural catheters in malignant effusions, there is a paucity of data regarding the use of ITPC in liver disease for the treatment of hepatic hydrothorax.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an indwelling tunneled pleural catheter (ITPC) in the management of hepatic hydrothorax that is not responsive to conventional medical therapy. Hepatic Hydrothorax (HH) is defined as an accumulation of fluid in the pleural space between the chest wall and the lung and occurs in 5-10% of patients with liver disease. Despite medical therapy with diuretics and salt restriction, many patients still experience intractable, debilitating shortness of breath, often necessitating hospital admission. Repeated thoracentesis,which is a procedure in which the hepatic hydrothorax is drained with a needle may be effective, but is often only temporary prior to the reaccumulation of fluid leading to the requirement of repeated procedures. Trans-jugular intrahepatic porto-systemic shunt (TIPS), while a valuable treatment for HH, is not always effective or able to be performed. Similarly, liver transplantation although potentially curative, is not available to many patients and may be significantly delayed. Many patients do not experience sufficient or timely relief with current conventional therapy.

DETAILED DESCRIPTION:
Hepatic Hydrothorax (HH) occurs in 5-10% of cirrhotic patients and remains a significant clinical challenge. Despite medical therapy with diuretics and sodium restriction, many patients still experience intractable, debilitating dyspnea and respiratory compromise. Repeated thoracentesis, while often effective, may affect prohibitively transient symptom relief and exposes the patient to repeated procedures with inherent cumulative risk. Trans-jugular intrahepatic porto-systemic shunt (TIPS), while a valuable treatment for HH, is not always effective or able to be performed. Similarly, liver transplantation although potentially curative, is not available to many patients and may be significantly delayed. Many patients do not experience sufficient or timely relief with current conventional therapy. There exists the need for additional therapies, either as a bridge to transplantation or TIPS, or for palliation when transplantation is not expected.

The insertion of an Indwelling tunneled pleural catheters (ITPC) may prove to be safe and effective in treating the dyspnea, cough, and hypoxemia associated with HH in patients refractory to conventional medical management, and serve as an effective bridge to transplantation or TIPS.

ITPCs have been shown to successfully and safely control dyspnea in patients with malignant pleural effusions; producing long-lasting plurodesis in greater than 50% of recipients. Compared to the large amount of published data regarding the use of ITPC in malignant effusions, there is a paucity of data regarding the use of ITPC in benign disease; particularly HH. A small series of four patients and a single case report have previously described the successful use of an ITPC for the management of HH. There exists the need for a prospective study to investigate the potential benefit of using ITPCs in patients with HH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have recurrent pleural effusion due to underlying cirrhosis
* Subjects who are potential candidates for liver transplantation
* Subjects who are candidates for transjugular intrahepatic portosystemic shunt procedures
* Subjects who have had at least one thoracentesis in the past three months

Exclusion Criteria:

* Subjects with active bacterial or fungal infection
* Subjectswho are not potential candidates for transplantation
* Subjects with pleural effusions due to processes other than cirrhosis
* Subjects who are critically ill at the time of referral, requiring intensive care unit admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2015-07-20 (Actual); Study Completion 2015-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Universtiy, St Louis, Missouri, United States

REFERENCES:
- [Derived] Chen A, Massoni J, Jung D, Crippin J. Indwelling Tunneled Pleural Catheters for the Management of Hepatic Hydrothorax. A Pilot Study. Ann Am Thorac Soc. 2016 Jun;13(6):862-6. doi: 10.1513/AnnalsATS.201510-688BC. PMID 27015392

RESULTS

PARTICIPANT FLOW:
Groups:
- ITPC: Patients in the ITPC (indwelling tunneled pleural catheter) arm will consist of patients with hepatic hydrothorax who have undergone at least one prior thoracentesis which has resulted in improvement in shortness of breath. The fluid characteristics will be consistent with a transudative pleural effusion. Patients in this group will also have been assessed by the Hepatology service and deemed candidates for additional therapy, such as liver transplant, or TIPS (transjugular intrahepatic portosystemic shunt).
Period: Overall Study
Arm/Group | ITPC
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ITPC: Patients in the ITPC (indwelling tunneled pleural catheter) arm will have and ITPC placed for management of recurrent pleural effusion due to liver disease (hepatic hydrothorax). These patients will have undergone at least one prior thoracentesis that has resulted in improvement in shortness of breath. Pleural fluid studies will demonstrate a transudative process, also consistent with hepatic hydrothorax. All patients will have undergone evaluation by the Hepatology service and will have been deemed eligible for additional treatment, such as liver transplant or TIPS (transjugular intrahepatic portosystemic shunt) procedures.
Arm/Group | ITPC
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Using Indwelling Tunneled Pleural Catheters for the Management of Hepatic Hydrothorax
Description: Feasibility of using ITPC's for the management of hepatic hydrothorax was assessed by the ability of patients to drain pleural effusions routinely via an indwelling tunneled pleural catheter for control of dyspnea related to pleural fluid accumulation. Feasibility was defined as successful catheter placement and improvement in shortness of breath following the procedure. Shortness of breath measurement was descriptive and self reported by patients on routine clinical follow up. Feasibility was also defined as patient ability to drain pleural effusions routinely at home. This was documented by patient logs documenting drainage.
Time Frame: From date of ITPC administration until the date of first documented complication such as infection that would require catheter removal or date of pleurodesis, whichever came first, assessed up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ITPC
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Arm/Group | ITPC
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No